CLINICAL TRIAL: NCT06173570
Title: A Phase IIb, Multicenter, Randomized, Parallel-Group, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy, Safety, and Tolerability of AZD0780 in Participants With Dyslipidemia
Brief Title: A Study to Assess the Efficacy, Safety and Tolerability of Different Doses of AZD0780 in Patients With Dyslipidemia
Acronym: PURSUIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7960C00006; 2023-506197-12-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-12-08; First posted 2023-12-15 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Dyslipidemia
Keywords: Dyslipidemia,; Low-Density Lipoprotein Cholesterol
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Intervention Model Description: Participants will be randomized with equal distribution across 5 parallel treatment arms to either placebo or one of four AZD0780 doses.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A (Experimental): AZD0780, Dose 1
  Interventions: Drug: AZD0780
- Arm B (Experimental): AZD0780, Dose 2
  Interventions: Drug: AZD0780
- Arm C (Experimental): AZD0780, Dose 3
  Interventions: Drug: AZD0780
- Arm D (Experimental): AZD0780, Dose 4
  Interventions: Drug: AZD0780
- Arm E (Placebo Comparator): Placebo, matched for appearance
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD0780 — AZD0780 administered orally, once daily for 12 weeks
  Arms: Arm A; Arm B; Arm C; Arm D
Drug: Placebo — Placebo administered orally, once daily for 12 weeks
  Arms: Arm E

SUMMARY:
The primary purpose of this study is to measure the effect of different daily doses of AZD0780 on Low-Density Lipoprotein (LDL-C) levels compared with placebo in participants with dyslipidemia. The effect of AZD0780 versus placebo on other lipid parameters and inflammatory markers is also investigated. The concentration of AZD0780 in blood at specific timepoints is measured, and the safety and tolerability of AZD0780 will be evaluated. There is a follow-up after end of treatment, but expanded access is not available. The primary hypothesis is that at least one of the investigated doses of AZD0780 is superior to placebo in lowering LDL-C level, in percent change from baseline up to week 12.

ELIGIBILITY:
Inclusion Criteria:

* Males, and females of non-childbearing potential 18 to 75 years of age, inclusive, at the time of signing the informed consent.
* Participants with a fasting low-density lipoprotein cholesterol (LDL-C) higher than or equal to 70 mg/dL (1.8 mmol/L) and lower than 190 mg/dL (4.9 mmol/L) at screening.
* Participants with fasting triglycerides lower than 400 mg/dL (lower than 4.52 mmol/L) at screening.
* Should be receiving moderate or high-intensity statin therapy for more than or equal to 2 months prior to screening.
* There should be no planned medication or dose change during study participation.
* Body mass index at or above 19.0 kg/m^2.

Exclusion Criteria:

* History or presence of gastrointestinal, hepatic or renal disease or any other conditions known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any uncontrolled or serious disease, or any medical (e.g., known major active infection or major hematological, renal, metabolic, gastrointestinal, respiratory, or endocrine dysfunction) or surgical condition that, in the opinion of the investigator, may either interfere with participation in the clinical study and/or put the participant at significant risk.
* Poorly controlled type 2 diabetes mellitus, defined as hemoglobin A1c (HbA1c) greater than 10 percent at screening.
* Acute ischemic cardiovascular event in the last 12 months.
* Heart failure with New York Heart Association (NYHA) Class III-IV.
* Malignancy (except non-melanoma skin cancers, cervical in-situ carcinoma, breast ductal carcinoma in-situ, or Stage 1 prostate carcinoma) within the last 10 years.
* Recipient of any major organ transplant, e.g., lung, liver, heart, bone marrow, renal.
* LDL or plasma apheresis within 12 months prior to randomization.
* Uncontrolled hypertension.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12 lead ECG as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (14):
  - Research Site, Huntsville, Alabama
  - Research Site, Lincoln, California
  - Research Site, Palm Springs, California
  - Research Site, Santa Ana, California
  - Research Site, Boca Raton, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Inverness, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, New Windsor, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, San Marcos, Texas
- Canada (6):
  - Research Site, Barrie, Ontario
  - Research Site, Brampton, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Concord, Ontario
  - Research Site, Guelph, Ontario
  - Research Site, Toronto, Ontario
- Czechia (9):
  - Research Site, Benešov
  - Research Site, Brandýs nad Labem
  - Research Site, Brno
  - Research Site, Louny
  - Research Site, Náchod
  - Research Site, Prague
  - Research Site, Příbram
  - Research Site, Teplice
  - Research Site, Uherské Hradiště
- Denmark (5):
  - Research Site, Aarhus
  - Research Site, Herning
  - Research Site, Hvidovre
  - Research Site, Svendborg
  - Research Site, Viborg
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Orosháza
  - Research Site, Pécs
- Japan (2):
  - Research Site, Chūōku
  - Research Site, Itabashi-ku
- Slovakia (7):
  - Research Site, Bratislava
  - Research Site, Brezno
  - Research Site, Lučenec
  - Research Site, Prešov
  - Research Site, Rožňava
  - Research Site, Svidník
  - Research Site, Trebišov
- Spain (6):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Ferrol
  - Research Site, Santiago(A Coruña)
  - Research Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Koren MJ, Vega RB, Agrawal N, Xu Y, Barbour AM, Yu H, Wallerstedt E, Carter D, Middlemiss J, Twaddle L, McCarthy MC, Rosenmeier JB. An Oral PCSK9 Inhibitor for Treatment of Hypercholesterolemia: The PURSUIT Randomized Trial. J Am Coll Cardiol. 2025 Jun 3;85(21):1996-2007. doi: 10.1016/j.jacc.2025.03.499. Epub 2025 Mar 31. PMID 40167413
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7960C00006&attachmentIdentifier=508a78db-c5c4-402d-81b5-83753173af0f&fileName=D7960C00006_Redacted_CSP.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7960C00006&attachmentIdentifier=6e6b323a-5a59-4b2d-b988-64464a1a5665&fileName=D7960C00006_Redacted_SAP.pdf&versionIdentifier=
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7960C00006&attachmentIdentifier=41bf0094-961d-4ca7-ab8d-9d108d244d58&fileName=D7960C00006_Redacted_CSR_Synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from January 2024 to September 2024 in 55 research sites in 8 countries (United States, Canada, Czech Republic, Denmark, Hungary, Japan, Slovakia, and Spain).
Pre-assignment Details: Of 428 enrolled participants, two randomized participants - one screen failure and one withdrawal by subject - did not start treatment.
Groups:
- AZD0780 1 mg: Participants received 1 mg of AZD0780 administered orally once daily for up to 12 weeks
- AZD0780 3 mg: Participants received 3 mg of AZD0780 administered orally once daily for up to 12 weeks
- AZD0780 10 mg: Participants received 10 mg of AZD0780 administered orally once daily for up to 12 weeks
- AZD0780 30 mg: Participants received 30 mg of AZD0780 administered orally once daily for up to 12 weeks
- Placebo: Participants received placebo administered orally once daily for up to 12 weeks
Period: Overall Study
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Started | 86 | 85 | 85 | 85 | 87
Started Treatment | 86 | 85 | 84 | 85 | 86
Completed | 81 | 81 | 84 | 80 | 82
Not Completed | 5 | 4 | 1 | 5 | 5
Not completed — Adverse Event | 1 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 1
Not completed — Non-compliance with Study Drug | 1 | 0 | 0 | 0 | 0
Not completed — Screen Failure | 0 | 0 | 0 | 0 | 1
Not completed — Other | 2 | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo | Total
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86 | 426
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 47 | 59 | 39 | 50 | 47 | 242
  >=65 years | 39 | 26 | 45 | 35 | 39 | 184
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (7.9) | 60.9 (7.2) | 63.9 (7.2) | 62.3 (7.9) | 62.3 (7.8) | 62.4 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 37 | 41 | 44 | 204
  Male | 45 | 44 | 47 | 44 | 42 | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 10 | 6 | 12 | 8 | 41
  Not Hispanic or Latino | 81 | 75 | 78 | 73 | 78 | 385
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 8 | 6 | 6 | 6 | 6 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 4 | 4 | 6 | 22
  White | 73 | 75 | 73 | 74 | 73 | 368
  More than one race | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 2
Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mmol/L] | 2.6822 (0.6918) | 2.7258 (0.8960) | 2.4784 (0.7122) | 2.5500 (0.6939) | 2.5769 (0.6620) | 2.6031 (0.7378)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) Level From Baseline to Week 12
Description: Percent change was calculated as (Week 12 LDL-C - Baseline LDL-C) / Baseline LDL-C * 100. Negative values indicate reduction in LDL-C. Baseline is the last non-missing value prior to first administration of study treatment. Hypothetical estimand: data collected after intercurrent events (ICEs) defined in the CSP excluded.
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86
Percent Change (%) | -31.19 [-37.06 to -25.32] | -33.83 [-39.78 to -27.88] | -41.09 [-46.92 to -35.25] | -46.62 [-52.48 to -40.76] | 4.08 [-1.84 to 10.00]
Statistical Analysis 1: Comparison: AZD0780 1 mg vs Placebo; MMRM with fixed effects for baseline LDL-C, treatment, visit, treatment-by-visit; random intercept for participants. Missing Week 12 LDL-C values handled by the MMRM under MAR. Hierarchical testing (in the order of decreasing dose of study treatment) controls two-sided alpha = 0.05; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -35.27, 95% CI 2-sided [-43.61 to -26.93] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 2: Comparison: AZD0780 3 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -37.91, 95% CI 2-sided [-46.31 to -29.51] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 3: Comparison: AZD0780 10 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -45.17, 95% CI 2-sided [-53.47 to -36.86] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 4: Comparison: AZD0780 30 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -50.70, 95% CI 2-sided [-59.03 to -42.37] — Difference = AZD0780 - Placebo; negative values favor AZD0780

2. Secondary Outcome: Percent Change From Baseline of Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12
Description: Percent change was calculated as (Week 12 LDL-C - Baseline LDL-C) / Baseline LDL-C * 100. Negative values indicate reduction in LDL-C. Baseline is the last non-missing value prior to first administration of study treatment. Treatment policy estimand: data collected after ICEs defined in the CSP retained.
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86
Percent Change (%) | -30.47 [-36.45 to -24.49] | -33.35 [-39.44 to -27.26] | -40.47 [-46.42 to -34.53] | -46.41 [-52.48 to -40.35] | 3.39 [-2.63 to 9.40]
Statistical Analysis 1: Comparison: AZD0780 1 mg vs Placebo; MMRM with fixed effects for baseline LDL-C, treatment, visit, treatment-by-visit; random intercept for participants. Missing data imputed using multiple imputation approach detailed in SAP Appendix 7.1; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -33.85, 95% CI 2-sided [-42.34 to -25.37] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 2: Comparison: AZD0780 3 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -36.73, 95% CI 2-sided [-45.30 to -28.17] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 3: Comparison: AZD0780 10 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -43.86, 95% CI 2-sided [-52.31 to -35.41] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 4: Comparison: AZD0780 30 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -49.80, 95% CI 2-sided [-58.35 to -41.25] — Difference = AZD0780 - Placebo; negative values favor AZD0780

3. Secondary Outcome: Percent Change From Baseline of Total Cholesterol at Week 12
Description: Percent change was calculated as (Week 12 value - Baseline value) / Baseline value * 100. Negative values indicate reduction in lipid parameter. Baseline is the last non-missing value prior to first administration of study treatment. Hypothetical estimand: data collected after intercurrent events (ICEs) defined in the CSP excluded.
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86
Percent Change (%) | -18.93 [-22.48 to -15.38] | -20.09 [-23.70 to -16.48] | -24.84 [-28.36 to -21.32] | -27.06 [-30.62 to -23.51] | 2.29 [-1.29 to 5.88]
Statistical Analysis 1: Comparison: AZD0780 1 mg vs Placebo; MMRM with fixed effects for baseline of the respective parameter, treatment, visit, treatment-by-visit; random intercept for participants. Missing Week 12 values handled by the MMRM under MAR; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -21.22, 95% CI 2-sided [-26.27 to -16.18] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 2: Comparison: AZD0780 3 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -22.39, 95% CI 2-sided [-27.48 to -17.30] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 3: Comparison: AZD0780 10 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -27.14, 95% CI 2-sided [-32.16 to -22.11] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 4: Comparison: AZD0780 30 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -29.36, 95% CI 2-sided [-34.40 to -24.31] — Difference = AZD0780 - Placebo; negative values favor AZD0780

4. Secondary Outcome: Percent Change From Baseline of High-Density Lipoprotein Cholesterol (HDL-C) at Week 12
Description: as for outcome 3
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86
Percent Change (%) | 0.12 [-2.96 to 3.19] | 4.03 [0.93 to 7.12] | 1.97 [-1.07 to 5.00] | 4.66 [1.60 to 7.72] | 3.65 [0.58 to 6.71]
Statistical Analysis 1: Comparison: AZD0780 1 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.111, Mixed Models Analysis; Mean Difference (Net) = -3.53, 95% CI 2-sided [-7.87 to 0.81] — Difference = AZD0780 - Placebo; positive values favor AZD0780
Statistical Analysis 2: Comparison: AZD0780 3 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.864, Mixed Models Analysis; Mean Difference (Net) = 0.38, 95% CI 2-sided [-3.98 to 4.74] — Difference = AZD0780 - Placebo; positive values favor AZD0780
Statistical Analysis 3: Comparison: AZD0780 10 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.445, Mixed Models Analysis; Mean Difference (Net) = -1.68, 95% CI 2-sided [-5.99 to 2.63] — Difference = AZD0780 - Placebo; positive values favor AZD0780
Statistical Analysis 4: Comparison: AZD0780 30 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.648, Mixed Models Analysis; Mean Difference (Net) = 1.01, 95% CI 2-sided [-3.32 to 5.34] — Difference = AZD0780 - Placebo; positive values favor AZD0780

5. Secondary Outcome: Percent Change From Baseline of Triglycerides at Week 12
Description: as for outcome 3
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86
Percent Change (%) | 3.06 [-5.05 to 11.17] | 2.90 [-5.29 to 11.08] | 1.93 [-5.99 to 9.85] | -0.44 [-8.52 to 7.63] | 9.56 [1.47 to 17.65]
Statistical Analysis 1: Comparison: AZD0780 1 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.266, Mixed Models Analysis; Mean Difference (Net) = -6.50, 95% CI 2-sided [-17.97 to 4.96] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 2: Comparison: AZD0780 3 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.256, Mixed Models Analysis; Mean Difference (Net) = -6.67, 95% CI 2-sided [-18.17 to 4.84] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 3: Comparison: AZD0780 10 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.186, Mixed Models Analysis; Mean Difference (Net) = -7.63, 95% CI 2-sided [-18.95 to 3.69] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 4: Comparison: AZD0780 30 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.086, Mixed Models Analysis; Mean Difference (Net) = -10.00, 95% CI 2-sided [-21.44 to 1.43] — Difference = AZD0780 - Placebo; negative values favor AZD0780

6. Secondary Outcome: Percent Change From Baseline of Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) at Week 12
Description: as for outcome 3
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86
Percent Change (%) | -26.85 [-32.65 to -21.04] | -29.86 [-35.75 to -23.97] | -35.13 [-40.92 to -29.35] | -41.65 [-47.45 to -35.85] | 3.53 [-2.33 to 9.39]
Statistical Analysis 1: Comparison: AZD0780 1 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -30.38, 95% CI 2-sided [-38.63 to -22.12] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 2: Comparison: AZD0780 3 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -33.39, 95% CI 2-sided [-41.71 to -25.08] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 3: Comparison: AZD0780 10 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -38.66, 95% CI 2-sided [-46.90 to -30.43] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 4: Comparison: AZD0780 30 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -45.18, 95% CI 2-sided [-53.43 to -36.94] — Difference = AZD0780 - Placebo; negative values favor AZD0780

7. Secondary Outcome: Percent Change From Baseline of Very-Low-Density Lipoprotein Cholesterol (VLDL-C) at Week 12
Description: as for outcome 3
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86
Percent Change (%) | 1.13 [-6.55 to 8.81] | 4.02 [-3.69 to 11.73] | 2.21 [-5.26 to 9.68] | 0.46 [-7.15 to 8.07] | 7.19 [-0.52 to 14.90]
Statistical Analysis 1: Comparison: AZD0780 1 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.276, Mixed Models Analysis; Mean Difference (Net) = -6.06, 95% CI 2-sided [-16.96 to 4.84] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 2: Comparison: AZD0780 3 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.568, Mixed Models Analysis; Mean Difference (Net) = -3.17, 95% CI 2-sided [-14.08 to 7.73] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 3: Comparison: AZD0780 10 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.363, Mixed Models Analysis; Mean Difference (Net) = -4.98, 95% CI 2-sided [-15.71 to 5.75] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 4: Comparison: AZD0780 30 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.223, Mixed Models Analysis; Mean Difference (Net) = -6.73, 95% CI 2-sided [-17.57 to 4.11] — Difference = AZD0780 - Placebo; negative values favor AZD0780

8. Secondary Outcome: Percent Change From Baseline of Apolipoprotein A1 at Week 12
Description: as for outcome 3
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86
Percent Change (%) | 1.67 [-1.00 to 4.34] | 3.25 [0.58 to 5.93] | 3.61 [1.02 to 6.21] | 5.72 [3.08 to 8.36] | 4.46 [1.80 to 7.12]
Statistical Analysis 1: Comparison: AZD0780 1 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.146, Mixed Models Analysis; Mean Difference (Net) = -2.79, 95% CI 2-sided [-6.56 to 0.98] — Difference = AZD0780 - Placebo; positive values favor AZD0780
Statistical Analysis 2: Comparison: AZD0780 3 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.530, Mixed Models Analysis; Mean Difference (Net) = -1.21, 95% CI 2-sided [-4.98 to 2.56] — Difference = AZD0780 - Placebo; positive values favor AZD0780
Statistical Analysis 3: Comparison: AZD0780 10 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.654, Mixed Models Analysis; Mean Difference (Net) = -0.85, 95% CI 2-sided [-4.56 to 2.87] — Difference = AZD0780 - Placebo; positive values favor AZD0780
Statistical Analysis 4: Comparison: AZD0780 30 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.509, Mixed Models Analysis; Mean Difference (Net) = 1.26, 95% CI 2-sided [-2.48 to 5.00] — Difference = AZD0780 - Placebo; positive values favor AZD0780

9. Secondary Outcome: Percent Change From Baseline of Apolipoprotein B at Week 12
Description: as for outcome 3
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86
Percent Change (%) | -24.08 [-28.37 to -19.80] | -25.39 [-29.71 to -21.07] | -34.33 [-38.53 to -30.12] | -36.95 [-41.20 to -32.71] | 2.92 [-1.39 to 7.23]
Statistical Analysis 1: Comparison: AZD0780 1 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -27.00, 95% CI 2-sided [-33.08 to -20.93] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 2: Comparison: AZD0780 3 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -28.31, 95% CI 2-sided [-34.42 to -22.20] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 3: Comparison: AZD0780 10 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -37.25, 95% CI 2-sided [-43.27 to -31.23] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 4: Comparison: AZD0780 30 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -39.87, 95% CI 2-sided [-45.92 to -33.83] — Difference = AZD0780 - Placebo; negative values favor AZD0780

10. Secondary Outcome: Percent Change From Baseline of Total Cholesterol at Week 12
Description: Percent change was calculated as (Week 12 value - Baseline value) / Baseline value * 100. Negative values indicate reduction in lipid parameter. Baseline is the last non-missing value prior to first administration of study treatment. Treatment policy estimand: data collected after ICEs defined in the CSP retained.
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86
Percent Change (%) | -18.23 [-21.88 to -14.58] | -19.80 [-23.54 to -16.07] | -24.54 [-28.14 to -20.94] | -26.90 [-30.60 to -23.20] | 1.73 [-1.88 to 5.34]
Statistical Analysis 1: Comparison: AZD0780 1 mg vs Placebo; MMRM with fixed effects for baseline of the respective parameter, treatment, visit, treatment-by-visit; random intercept for participants. Missing data imputed using multiple imputation approach detailed in SAP Appendix 7.1; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -19.96, 95% CI 2-sided [-25.09 to -14.84] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 2: Comparison: AZD0780 3 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -21.54, 95% CI 2-sided [-26.73 to -16.35] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 3: Comparison: AZD0780 10 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -26.27, 95% CI 2-sided [-31.37 to -21.18] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 4: Comparison: AZD0780 30 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -28.64, 95% CI 2-sided [-33.80 to -23.48] — Difference = AZD0780 - Placebo; negative values favor AZD0780

11. Secondary Outcome: Percent Change From Baseline of High-Density Lipoprotein Cholesterol (HDL-C) at Week 12
Description: as for outcome 10
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86
Percent Change (%) | 0.80 [-2.29 to 3.89] | 3.66 [0.58 to 6.75] | 2.17 [-0.85 to 5.19] | 4.65 [1.61 to 7.70] | 3.11 [0.11 to 6.12]
Statistical Analysis 1: Comparison: AZD0780 1 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.292, Mixed Models Analysis; Mean Difference (Net) = -2.31, 95% CI 2-sided [-6.62 to 1.99] — Difference = AZD0780 - Placebo; positive values favor AZD0780
Statistical Analysis 2: Comparison: AZD0780 3 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.802, Mixed Models Analysis; Mean Difference (Net) = 0.55, 95% CI 2-sided [-3.76 to 4.86] — Difference = AZD0780 - Placebo; positive values favor AZD0780
Statistical Analysis 3: Comparison: AZD0780 10 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.664, Mixed Models Analysis; Mean Difference (Net) = -0.94, 95% CI 2-sided [-5.21 to 3.32] — Difference = AZD0780 - Placebo; positive values favor AZD0780
Statistical Analysis 4: Comparison: AZD0780 30 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.481, Mixed Models Analysis; Mean Difference (Net) = 1.54, 95% CI 2-sided [-2.74 to 5.82] — Difference = AZD0780 - Placebo; positive values favor AZD0780

12. Secondary Outcome: Percent Change From Baseline of Triglycerides at Week 12
Description: as for outcome 10
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86
Percent Change (%) | 2.81 [-5.25 to 10.86] | 2.17 [-5.93 to 10.28] | 1.72 [-6.09 to 9.54] | -0.83 [-8.87 to 7.22] | 9.04 [1.16 to 16.92]
Statistical Analysis 1: Comparison: AZD0780 1 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.278, Mixed Models Analysis; Mean Difference (Net) = -6.23, 95% CI 2-sided [-17.50 to 5.03] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 2: Comparison: AZD0780 3 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.234, Mixed Models Analysis; Mean Difference (Net) = -6.87, 95% CI 2-sided [-18.19 to 4.45] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 3: Comparison: AZD0780 10 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.196, Mixed Models Analysis; Mean Difference (Net) = -7.32, 95% CI 2-sided [-18.41 to 3.78] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 4: Comparison: AZD0780 30 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.086, Mixed Models Analysis; Mean Difference (Net) = -9.87, 95% CI 2-sided [-21.14 to 1.41] — Difference = AZD0780 - Placebo; negative values favor AZD0780

13. Secondary Outcome: Percent Change From Baseline of Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) at Week 12
Description: as for outcome 10
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86
Percent Change (%) | -26.13 [-31.94 to -20.32] | -29.42 [-35.34 to -23.49] | -34.77 [-40.59 to -28.95] | -41.35 [-47.27 to -35.43] | 2.86 [-2.91 to 8.62]
Statistical Analysis 1: Comparison: AZD0780 1 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -28.99, 95% CI 2-sided [-37.16 to -20.81] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 2: Comparison: AZD0780 3 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -32.28, 95% CI 2-sided [-40.54 to -24.02] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 3: Comparison: AZD0780 10 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -37.63, 95% CI 2-sided [-45.82 to -29.44] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 4: Comparison: AZD0780 30 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -44.21, 95% CI 2-sided [-52.47 to -35.94] — Difference = AZD0780 - Placebo; negative values favor AZD0780

14. Secondary Outcome: Percent Change From Baseline of Very-Low-Density Lipoprotein Cholesterol (VLDL-C) at Week 12
Description: as for outcome 10
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86
Percent Change (%) | 0.81 [-6.81 to 8.43] | 2.67 [-4.91 to 10.26] | 1.77 [-5.59 to 9.13] | 0.42 [-7.18 to 8.02] | 6.74 [-0.68 to 14.15]
Statistical Analysis 1: Comparison: AZD0780 1 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.275, Mixed Models Analysis; Mean Difference (Net) = -5.93, 95% CI 2-sided [-16.57 to 4.71] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 2: Comparison: AZD0780 3 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.451, Mixed Models Analysis; Mean Difference (Net) = -4.06, 95% CI 2-sided [-14.63 to 6.51] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 3: Comparison: AZD0780 10 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.351, Mixed Models Analysis; Mean Difference (Net) = -4.97, 95% CI 2-sided [-15.41 to 5.47] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 4: Comparison: AZD0780 30 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.243, Mixed Models Analysis; Mean Difference (Net) = -6.32, 95% CI 2-sided [-16.92 to 4.29] — Difference = AZD0780 - Placebo; negative values favor AZD0780

15. Secondary Outcome: Percent Change From Baseline of Apolipoprotein A1 at Week 12
Description: as for outcome 10
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86
Percent Change (%) | 2.52 [-0.18 to 5.22] | 2.89 [0.14 to 5.64] | 3.79 [1.19 to 6.39] | 5.55 [2.88 to 8.22] | 3.82 [1.15 to 6.48]
Statistical Analysis 1: Comparison: AZD0780 1 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.501, Mixed Models Analysis; Mean Difference (Net) = -1.30, 95% CI 2-sided [-5.08 to 2.48] — Difference = AZD0780 - Placebo; positive values favor AZD0780
Statistical Analysis 2: Comparison: AZD0780 3 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.634, Mixed Models Analysis; Mean Difference (Net) = -0.93, 95% CI 2-sided [-4.74 to 2.89] — Difference = AZD0780 - Placebo; positive values favor AZD0780
Statistical Analysis 3: Comparison: AZD0780 10 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.990, Mixed Models Analysis; Mean Difference (Net) = -0.02, 95% CI 2-sided [-3.74 to 3.70] — Difference = AZD0780 - Placebo; positive values favor AZD0780
Statistical Analysis 4: Comparison: AZD0780 30 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.366, Mixed Models Analysis; Mean Difference (Net) = 1.73, 95% CI 2-sided [-2.03 to 5.50] — Difference = AZD0780 - Placebo; positive values favor AZD0780

16. Secondary Outcome: Percent Change From Baseline of Apolipoprotein B at Week 12
Description: as for outcome 10
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 86 | 85 | 84 | 85 | 86
Percent Change (%) | -23.35 [-27.79 to -18.91] | -24.53 [-29.06 to -19.99] | -33.85 [-38.18 to -29.51] | -36.86 [-41.35 to -32.37] | 2.44 [-2.00 to 6.89]
Statistical Analysis 1: Comparison: AZD0780 1 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -25.79, 95% CI 2-sided [-32.08 to -19.51] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 2: Comparison: AZD0780 3 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -26.97, 95% CI 2-sided [-33.33 to -20.62] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 3: Comparison: AZD0780 10 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -36.29, 95% CI 2-sided [-42.50 to -30.08] — Difference = AZD0780 - Placebo; negative values favor AZD0780
Statistical Analysis 4: Comparison: AZD0780 30 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -39.30, 95% CI 2-sided [-45.61 to -32.99] — Difference = AZD0780 - Placebo; negative values favor AZD0780

17. Secondary Outcome: Percent Change From Baseline of Lipoprotein-a at Week 12
Description: Percent change was calculated as (Week 12 value - Baseline value) / Baseline value * 100. Negative values indicate reduction in lipid parameter. Baseline is the last non-missing value prior to first administration of study treatment. Descriptive statistics only.
Time Frame: From first day of treatment up to week 12
Population: Full Analysis Set: all randomized participants who received at least one dose of study treatment. For this outcome, only participants with both baseline and week 12 values were included in the analysis.
Measure: Median (Full Range); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 75 | 75 | 81 | 76 | 78
Percent Change (%) | -7.48 [-64.6 to 319.6] | -11.16 [-56.7 to 2582.3] | -19.57 [-66.3 to 36.6] | -19.43 [-71.3 to 55.6] | 0.00 [-46.3 to 98.9]

18. Secondary Outcome: Percent Change From Baseline of Remnant Cholesterol at Week 12
Description: as for outcome 17
Time Frame: From first day of treatment up to week 12
Population: as for outcome 17
Measure: Median (Full Range); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 75 | 75 | 79 | 77 | 80
Percent Change (%) | -9.09 [-77.8 to 160.0] | -8.33 [-169.7 to 671.4] | -22.95 [-1200.0 to 266.7] | -18.31 [-200.0 to 420.0] | -5.00 [-85.7 to 558.3]

19. Secondary Outcome: Percent Change From Baseline of High Sensitivity C-reactive Protein (hsCRP) at Week 12
Description: as for outcome 17
Time Frame: From first day of treatment up to week 12
Population: as for outcome 17
Measure: Median (Full Range); unit: Percent Change (%)
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
Number analyzed (Participants) | 75 | 75 | 82 | 77 | 79
Percent Change (%) | 0.00 [-96.8 to 2500.0] | 0.00 [-79.8 to 716.7] | 0.00 [-98.1 to 4950.0] | -22.22 [-93.3 to 2603.0] | 0.00 [-75.7 to 1358.3]

20. Secondary Outcome: AZD0780 Plasma Concentrations Summarized by Sampling Timepoint
Description: Geometric mean plasma concentration; LLOQ = 0.01 umol/L; BLQ values are handled as Not Quantified (NQ)
Time Frame: From week 1 up to week 12
Population: PK Analysis Set: all participants who received at least one dose of study treatment and who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: umol/L
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg
Number analyzed (Participants) | 85 | 83 | 84 | 84
umol/L
  Week 1: number analyzed (Participants) | 82 | 82 | 82 | 83
  Week 1 | 0.0790 (76.7603) | 0.2523 (54.0463) | 0.8120 (72.6051) | 2.6420 (58.0213)
  Week 2: number analyzed (Participants) | 84 | 83 | 82 | 84
  Week 2 | 0.0926 (71.7485) | 0.2639 (75.6804) | 0.8156 (95.1545) | 2.6676 (55.8538)
  Week 4: number analyzed (Participants) | 84 | 82 | 82 | 83
  Week 4 | 0.0901 (81.2970) | 0.2380 (98.8448) | 0.8393 (74.6636) | 2.7059 (47.5671)
  Week 8: number analyzed (Participants) | 80 | 82 | 83 | 81
  Week 8 | 0.0932 (68.6270) | 0.2359 (102.5351) | 0.8350 (92.9640) | 2.4911 (102.6420)
  Week 12: number analyzed (Participants) | 79 | 81 | 82 | 80
  Week 12 | 0.0957 (61.8573) | 0.2317 (111.2636) | 0.7221 (119.9436) | 2.4373 (134.1014)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of study treatment, throughout the 12-week treatment period, and the 2-weeks follow-up period.
Arm/Group | AZD0780 1 mg | AZD0780 3 mg | AZD0780 10 mg | AZD0780 30 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/85 | 0/84 | 0/85 | 0/86
Serious Adverse Events (participants affected / at risk) | 2/86 | 2/85 | 2/84 | 1/85 | 0/86
Other Adverse Events (participants affected / at risk) | 4/86 | 2/85 | 2/84 | 3/85 | 5/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD0780 1 mg (N=86) | AZD0780 3 mg (N=85) | AZD0780 10 mg (N=84) | AZD0780 30 mg (N=85) | Placebo (N=86)
Major Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD0780 1 mg (N=86) | AZD0780 3 mg (N=85) | AZD0780 10 mg (N=84) | AZD0780 30 mg (N=85) | Placebo (N=86)
Hypertension (Vascular disorders) | 4 (4) | 2 (2) | 2 (2) | 3 (3) | 5 (5)

LIMITATIONS AND CAVEATS:
The secondary endpoints - percent change from baseline in Lipoprotein-a, remnant cholesterol, and hsCRP at Week 12 - could not be reliably interpreted using the planned inferential statistics model due to individual unexpected values and skewed data. Therefore, the endpoint analyses use descriptive statistics to illustrate the data distribution for these parameters.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information may be disclosed without prior written approval from AstraZeneca AB.

DOCUMENTS (2):
  • Study Protocol (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT06173570/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT06173570/SAP_001.pdf